CLINICAL TRIAL: NCT06788509
Title: An Open Label, Rollover Platform Study for Continued Study Treatment and Ongoing Safety Monitoring
Brief Title: A Rollover Study for Continued Study Treatment and Ongoing Safety Monitoring
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLATFORMPACAN1001; PLATFORMPACAN1001 (Other: Janssen Research & Development, LLC); 2024-515457-21-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Neoplasms; Solid Tumor, Adult; Metastatic Castration-resistant Prostate Cancer (mCRPC)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes; Neoplasms | interventions — ibrutinib; JNJ-64264681; JNJ-64619178

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Long Term Safety Assessment (Platform Study) (Other): The platform rollover study provides continued long-term access to study treatment(s) (JNJ-64264681; JNJ-67856633 (safimaltib); JNJ-54179060 (ibrutinib); JNJ-75348780; JNJ-74856665; JNJ-64619178; JNJ-70218902) for participants currently receiving the active study treatment in parent studies and deriving benefit from it. Eligible participants in parent study will rollover to this platform study which will be adapted into Intervention Specific Appendix (ISA) within the platform study. Participants will initiate the platform study under the relevant ISA, and will continue to receive study treatment at the dose they received in parent study.
  Interventions: Drug: JNJ-75348780; Drug: JNJ-67856633; Drug: JNJ-54179060; Drug: JNJ-64264681; Drug: JNJ-74856665; Drug: JNJ-70218902; Drug: JNJ-64619178

INTERVENTIONS:
Drug: JNJ-75348780 — Participants from the parent study (75348780LYM1001 [NCT04540796]) who are deriving benefit from study treatment will continue to receive subcutaneous JNJ-75348780.
Drug: JNJ-67856633 — Participants from the parent studies (64264681LYM1002 [NCT04657224], 67856633LYM1002 [NCT04876092] and 67856633LYM1001 [NCT03900598]) who are deriving benefit from study treatment will continue to receive JNJ-67856633 orally.
  Other Names: safimaltib
Drug: JNJ-54179060 — Participants from the parent study (67856633LYM1002 [NCT04876092]) who are deriving benefit from study treatment will continue to receive JNJ-54179060 orally.
  Other Names: ibrutinib
Drug: JNJ-64264681 — Participants from the parent studies (64264681LYM1001 [NCT04210219], 64264681LYM1002 [NCT04657224]) who are deriving benefit from study treatment will continue to receive JNJ-64264681 orally.
Drug: JNJ-74856665 — Participants from the parent study (74856665AML1001 [NCT04609826]) who are deriving benefit from study treatment will continue to receive JNJ-74856665 orally.
Drug: JNJ-70218902 — Participants from the parent study (70218902EDI1001 [NCT04397276]) who are deriving benefit from study treatment will continue to receive JNJ-70218902 orally.
Drug: JNJ-64619178 — Participants from the parent study (64619178EDI1001 [NCT03573310]) who are deriving benefit from study treatment will continue to receive JNJ-64619178 orally.

SUMMARY:
The purpose of this study is to collect long-term safety data in participants with cancers including acute myeloid leukemia, non-Hodgkin lymphoma, myelodysplastic syndrome, chronic lymphocytic leukemia (type of cancer of the blood and bone marrow in which the bone marrow makes a large number of abnormal blood cells) and advanced solid tumors and metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Have participated in a parent study, with a linked intervention specific appendix (ISA) within this platform study, in which they initially received study treatment(s) prior to rolling over to this platform study
* Satisfy all ISA specific inclusion criteria
* Sign an informed consent form (ICF) (or their legally acceptable representative must sign) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the platform study with details per the relevant ISA
* Be willing and able to adhere to the lifestyle restrictions specified in the relevant ISA

Exclusion Criteria:

* Have any condition or situation which, in the opinion of the investigator, may put the subject at significant risk, may confound the study results, or may interfere significantly with subject's participation in the study
* Have unacceptable toxicities or overt disease progression observed at time of rollover to the respective ISA
* Meets any exclusion criteria within the pertinent ISA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2028-01-19 (Estimated); Study Completion 2028-01-21 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious Adverse Events (SAEs) and Grade Greater than or equals to (>=) 3 Related Adverse Events (AEs) | Up to approximately 3 years and 7 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the treatment. An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, is considered or defined as an important medical event, or abnormal pregnancy outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (26):
- Ghent University Hospital, Ghent, Belgium
- France (3):
  - Hopital Claude Huriez, Lille
  - CHU Nantes, Nantes
  - Institut Gustave Roussy, Villejuif
- Arensia Exploratory Medicine, Tbilisi, Georgia
- Alexandra Hospital, Athens, Greece
- Israel (2):
  - Rambam Medical Center, Haifa
  - Hadassah University Hospita Ein Kerem, Jerusalem
- Japan (2):
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - The Cancer Institute Hospital of JFCR, Tokyo
- Arensia Exploratory Medicine, Chisinau, Moldova
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne Osrodek Badan Klinicznych Wczesnych Faz, Gdansk
  - Pratia MCM Krakow, Krakow
  - Aidport Sp z o o, Skorzewo
- Severance Hospital Yonsei University Health System, Seoul, South Korea
- Spain (3):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
- Taiwan (4):
  - Chang Kung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Medical Center of Limited Liability Company Arensia Exploratory Medicine, Kyiv, Ukraine
- United Kingdom (3):
  - University Hospitals Of Leicester Nhs Trust, Leicester
  - St Bartholomews Hospital, London
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency